CLINICAL TRIAL: NCT04960397
Title: A Phase 1b, Double-Blind, Randomized, Dose-Escalating, Age De-Escalating, Placebo-Controlled Study to Assess the Safety and Immunogenicity of One or Two Doses of Sing2016 M2SR H3N2 Influenza Vaccine Delivered Intranasally In a Healthy Pediatric Population 6 Months Through 17 Years of Age.
Brief Title: Assess the Safety and Immunogenicity of One or Two Doses of Sing2016 M2SR H3N2 Influenza Vaccine
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Lack of product and funding.
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 20-0009; 75N93019C00055
Record Dates: First submitted 2021-07-08; First posted 2021-07-13 (Actual); Results first posted 2025-06-06 (Actual); Last update posted 2025-08-03 (Actual); Status verified 2025-04-18

CONDITIONS: H3N2 Influenza
Keywords: Healthy Pediatric Population; Immunogenicity; Influenza; M2SR H3N2 Influenza Vaccine; Phase 1b; Sing2016 M2SR H3N2 Influenza Vaccine
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Participants, site investigators, and study personnel performing any study-related assessments following study product administration are blinded to product received. Laboratory personnel performing immunological assays will receive serum blinded to participant ID number, specimen visit number, and allocation group.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Cohort 1 (Experimental): A cohort of influenza non-naïve 45 healthy children, 9-17 years old, will receive a single dose of 10^9 TCID50 of intranasal Sing2016 M2SR H3N2 vaccine (N=30) or placebo (N=15) at Day 1. N=45.
  Interventions: Other: Placebo; Biological: Sing2016 M2SR H3N2
- Cohort 2 (Experimental): A cohort of influenza non-naïve 45 healthy children, 2-8 years old, will receive a single dose of 10^8 TCID50 of intranasal Sing2016 M2SR H3N2 vaccine (N=30) or placebo (N=15) at Day 1 intranasally. N= 45
  Interventions: Other: Placebo; Biological: Sing2016 M2SR H3N2
- Cohort 3 (Experimental): Once, there is sufficient evidence of safety and tolerability in Cohorts 1 and 2,and enrollment has completed of all 45 in each of these cohorts. Cohort 3 will begin enrollment. A cohort of influenza non-naïve 25 healthy children, 2-8 years old, will receive a single dose of 10^9 TCID50 of intranasal Sing2016 M2SR H3N2 vaccine (N=15) or placebo (N=10) at Day 1. N=25.
  Interventions: Other: Placebo; Biological: Sing2016 M2SR H3N2
- Cohort 4 (Experimental): Once, there is sufficient evidence of safety and tolerability in Cohort 3 and enrollment has been completed for this cohort, and fifth cohorts (Cohorts 4 and 5) will begin enrollment. A cohort of influenza non-naïve 25 healthy children, 2-8 years old, will receive two doses of the 10^9 TCID50 of intranasal Sing2016 M2SR H3N2 vaccine (N=15) or two doses of placebo (N=10) at Day 1 and Day 29. N=25
  Interventions: Other: Placebo; Biological: Sing2016 M2SR H3N2

INTERVENTIONS:
Other: Placebo — Physiological saline, i.e., 0.9% sodium chloride.
Biological: Sing2016 M2SR H3N2 — Novel intranasal live attenuated influenza vaccine with a defective M2 gene which renders the virus unable to replicate and generate progeny in animals and in humans, making its infectivity self-limiting. It induces both a mucosal and cell-mediated immune response and is administered intranasally. Supplied by Flugen Inc.

SUMMARY:
This is a Phase 1b, randomized, double-blind, dose-escalating, age de-escalating, placebo-controlled study of 200 children, ages 6 months to 17 years. This clinical trial is designed to assess the safety, tolerability/reactogenicity, and immunogenicity of one and two doses of Sing2016 M2SR H3N2 influenza vaccine (manufactured by FluGen) administered intranasally in seven cohorts of children. The study design includes pre-planned Safety Review Committee( SRC) reviews.

The first two groups to be vaccinated will be Cohorts 1 and 2. Cohort 1 consists of 45 children 9-17 years old. Thirty of them will receive one dose of the vaccine at a dose of 10^9 TCID50, and 15 will receive one dose of placebo. Cohort 2 comprises 45 children 2-8 years old. Thirty of them will receive one dose of the vaccine at a dose of 10^8 TCID50 and 15 will receive one dose of placebo.

Cohort 3 consists of 25 children 2-8 years old. 15 of them will receive one dose of vaccine at 10^9 TCID50 and 10 will receive one dose of placebo. Once 25 participants in Cohort 3 have completed Day 8 of follow-up, similar to Cohorts 1 and 2, the SRC will review to ensure no halting rules are met and if no rules are met, and the SRC determines it is safe to proceed, simultaneous enrollment into Cohorts 4 and 5 can begin. If any halting rules are met or any concerns are raised by the SRC, an external SMC may meet to discuss the data for recommendations on either progression or clinical trial modification before progression to the next cohort.

Cohort 4 consists of 25 children 2-8 years old; 15 of them will receive two doses of vaccine at 10^9 TCID50 and 10 will receive two doses of placebo, with a 28-day interval between the first and second doses. Due to the limited availability of product, and funding to support additional years of enrollment into Cohorts 5, 6, and 7, the decision was made to stop enrollment after the final participant was enrolled into Cohort 4.

The primary study objective is to assess the safety and tolerability of one and two administrations of the Sing2016 M2SR H3N2 influenza vaccine at 10^8 or 10^9 TCID50 delivered intranasally to healthy participants, 2 to 17 years of age.

DETAILED DESCRIPTION:
This is a Phase 1b, randomized, double-blind, dose-escalating, age de-escalating, placebo-controlled study of 200 children, ages 6 months to 17 years. This clinical trial is designed to assess the safety, tolerability/reactogenicity, and immunogenicity of one and two doses of Sing2016 M2SR H3N2 influenza vaccine (manufactured by FluGen) administered intranasally in seven cohorts of children. The study design includes pre-planned Safety Review Committee( SRC) reviews.

The first two groups to be vaccinated will be Cohorts 1 and 2. Cohort 1 consists of 45 children 9-17 years old. Thirty of them will receive one dose of the vaccine at a dose of 10^9 TCID50, and 15 will receive one dose of placebo. Cohort 2 comprises 45 children 2-8 years old. Thirty of them will receive one dose of the vaccine at a dose of 10^8 TCID50 and 15 will receive one dose of placebo. Sites will enroll participants into Cohorts 1 and 2 simultaneously. Once 25 or more participants in each of the first 2 cohorts (Cohorts 1 and 2) have completed Day 8, SRC will evaluate if any halting rules are met and if it is deemed safe enrollment in Cohort 3 may open. Cohort 2 must fully enroll before enrollment in Cohort 3 may begin.

Cohort 3 consists of 25 children 2-8 years old. 15 of them will receive one dose of vaccine at 10^9 TCID50 and 10 will receive one dose of placebo. Once all 25 participants in Cohort 3 have completed Day 8 of follow-up, similar to Cohorts 1 and 2, the SRC will review to ensure no halting rules are met and if no rules are met, and the SRC determines it is safe to proceed, simultaneous enrollment into Cohorts 4 and 5 can begin. If any halting rules are met or any concerns are raised by the SRC, an external SMC may meet to discuss the data for recommendations on either progression or clinical trial modification before progression to the next cohort.

Cohort 4 consists of 25 children 2-8 years old; 15 of them will receive two doses of vaccine at 10^9 TCID50 and 10 will receive two doses of placebo, with a 28-day interval between the first and second doses. Due to the limited availability of product, and funding to support additional years of enrollment into Cohorts 5, 6, and 7, the decision was made to stop enrollment after the final participant was enrolled into Cohort 4.

The primary study objective is to assess the safety and tolerability of one and two administrations of the Sing2016 M2SR H3N2 influenza vaccine at 10^8 or 10^9 TCID50 delivered intranasally to healthy participants, 2 to 17 years of age. The secondary study objective is to assess the humoral immunogenicity (serum antibody and mucosal antibody responses) directed against homologous viral strains after one and two administrations of Sing2016 M2SR H3N2 influenza vaccine at 10^8 or 10^9 TCID50 delivered intranasally to healthy participants, 2 to 17 years of age.

ELIGIBILITY:
Inclusion Criteria:

1. Participant is a male or female child aged 6 months to 17 years inclusive at time of enrollment (each cohort has its own age upper and lower limits*)

* Cohort 1: 9-17 years (on or after the ninth birthday and before the eighteenth birthday at the time of the first dose); Cohorts 2, 3, and 4: 2-8 years (on or after the second birthday and before the ninth birthday at the time of the first dose); Cohorts 5, 6, and 7: 6 months to 23 months (on or after the sixth month of life based on calendar day and before the second birthday at the time of the first dose) 2. For Cohorts 1 to 4, receipt of at least 2 doses of seasonal influenza vaccine in the past.

  3. For Cohorts 5 to 7, receipt of no seasonal influenza vaccines in the past and no documented history of laboratory-confirmed influenza illness 4. Parent/guardian of the participating child provides written informed permission and participating child provides assent* prior to initiation of any study procedures
* As appropriate by age or development and approved by the Institutional Review Board (IRB) 5. Parent/guardian and participant, as appropriate, are able to understand and comply with planned study procedures and are available for all study visits 6. Participant is in good health as assessed by the principal investigator or other designated study investigator*
* Based on medical history and physical examination (physical examination may be done as part of routine medical care or specifically for eligibility screening) 7. Parent/guardian of the participating child agrees not to allow the participant to join another clinical trial that includes an investigational agent or device during the study period 8. A female participant of child-bearing potential* agrees to abstain from sexual intercourse or to correctly use an acceptable method of contraception**
* A female of child-bearing potential is defined as a female who is post-menarchal and not sterilized via tubal ligation, bilateral oophorectomy, salpingectomy, hysterectomy, or successful Essure (R) placement (permanent, non-surgical, non-hormonal sterilization) with documented radiological confirmation test at least 90 days after the procedure. This applies only to participants in Cohort 1.

  **Acceptable methods of contraception must be used from 30 days prior to vaccination until 60 days after the last study vaccination (not Inactivated Influenza Vaccine (IIV4)) and include full abstinence from sexual intercourse with a male partner, monogamous relationship with vasectomized partner who has been vasectomized for 180 days or more or shown to be azoospermic prior to the participant receiving the study vaccination, barrier methods such as condoms or diaphragms/cervical cap, intrauterine devices, NuvaRing (R), and licensed hormonal methods such as implants, injectables, or oral contraceptives ("the pill").

  9. A female participant of child-bearing potential must have a negative urine pregnancy test within 24 hours prior to each study product 10. A male who is sexually active with a female of childbearing potential must agree to use an acceptable method of contraception*
* From the time of the first dose of study vaccine until 60 days after receipt of the last dose study vaccine, only in cohort 1. The only acceptable method of contraception for males who are sexually active with females of childbearing potential is condoms.

Exclusion Criteria:

1. Has a body temperature of 38 degrees Celsius or 100.4 degrees Fahrenheit (oral or axillary) or greater or another acute illness* within the 72 hours prior to study vaccination

   *Potential participants who are recovering from an acute illness and have residual minimal symptoms, which, in the opinion of the site principal investigator or appropriate sub-investigator, will not likely affect the evaluation of outcome measures are not ineligible. Temperature evaluation will not be performed as a study procedure on participants prior to administration of seasonal influenza vaccine
2. Has any medical or mental health disease or condition* that would render study participation unsafe, or would interfere with the evaluation of the responses

   *In the opinion of the site principal investigator or appropriate sub-investigator
3. Has a history of provider-diagnosed asthma requiring the use of medications at any age or has had a wheezing episode or use of medications to treat asthma in the 12 months prior to screening.
4. Has immunosuppression as a result of an underlying illness or treatment, a recent history or current use of immunosuppressive or immunomodulating disease therapy
5. Has a diagnosis of or history of malignant neoplastic disease
6. Has taken oral, parenteral (intramuscular or intravenous), inhaled, or nasal corticosteroids of any dose within 30 days prior to study vaccination
7. Has known HIV, hepatitis B, or hepatitis C infection
8. Has known hypersensitivity or allergy to any components of the study vaccine or material in the nasal delivery device*

   *Vaccine components: sucrose, sodium chloride, phosphate, glutamate; delivery device material: polycarbonate, polypropylene, synthetic rubber
9. Has a history of severe reactions following previous immunization with licensed or unlicensed influenza vaccines
10. Has a history of an anatomic disorder of the nares or nasopharynx
11. Has a history of chronic sinus infections
12. Has a history of or currently smokes or vapes
13. Has a history of Guillain-Barré syndrome
14. Use of aspirin- or salicylate-containing products in the 30 days prior to or intends to use these products in the 30 days following administration of the investigational vaccine
15. Has a history of documented influenza or receipt of influenza antiviral treatment in the 4 months prior to the first vaccination
16. Receipt of any antiviral drug within the week prior to or following the investigational vaccine.
17. Receipt of a licensed live vaccine within 30 days prior to the first study vaccination or plans to receive a licensed live vaccine within the 30 days after the last study vaccination.
18. Receipt of licensed inactivated non-influenza vaccine within 14 days prior to the first study vaccination, or plans to receive licensed, inactivated vaccine within the 30 days after the last study vaccination. ** Participants will be asked to avoid receipt of any routine licensed vaccines or vaccines under emergency use authorization during the periods described.
19. Receipt of an influenza vaccine within the 4 months prior to the first study vaccination or plans to receive an influenza vaccine following the last study vaccination. Seasonal IIV4 will be received by participants as part of this trial.
20. Receipt of immunoglobulin or other blood products within the 6 months prior to the first study vaccination or plans to receive during the period of study participation.
21. Receipt of an experimental* agent or device within the 6 months prior to the first study vaccination or expects to receive an experimental agent or device during the study period.

    *Products for treatment or prevention of coronavirus disease 2019 (COVID-19), when received under Emergency Use Authorization (EUA) or full FDA approval and not as part of a clinical trial, will not be deemed "experimental" for the purposes of this criterion and will not make an otherwise eligible prospective participant ineligible.
22. Is a family member of study personnel or personnel directly involved in the conduct or monitoring of the study.
23. Receipt of an approved or experimental product for treatment or prevention of COVID-19 within the 10 days prior to study enrollment.

    * Participants may enroll if greater than 10 days after receipt of the COVID-19 treatment or prevention.
    * Participants who are receiving COVID-19 vaccines around the time of dosing of the investigational product will be asked to avoid COVID-19 vaccination within the 10 days before any vaccination in the study and within any reactogenicity period (the day of and 7 days following each intranasal vaccination).
24. Inability of the study team to collect 5 mL of blood from the participant before the first vaccination (pre-vaccination blood).

Ages: 6 Months to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 140 (Actual)
Dates: Start 2021-09-10 (Actual); Primary Completion 2024-04-12 (Actual); Study Completion 2024-04-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - University of Iowa - Infectious Disease Clinic, Iowa City, Iowa
  - University of Maryland, School of Medicine, Center for Vaccine Development and Global Health, Baltimore, Maryland
  - Duke Vaccine and Trials Unit, Durham, North Carolina
  - Vanderbilt University - Pediatric - Vanderbilt Vaccine Research Center, Nashville, Tennessee

REFERENCES:
- [Derived] Taaffe J, Ostrowsky JT, Mott J, Goldin S, Friede M, Gsell P, Chadwick C. Advancing influenza vaccines: A review of next-generation candidates and their potential for global health impact. Vaccine. 2024 Dec 2;42(26):126408. doi: 10.1016/j.vaccine.2024.126408. Epub 2024 Oct 5. PMID 39369576

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were healthy children (ages 2-17 years) meeting all protocol-defined eligibility criteria.
  Recruited between August 19, 2021 and September 15, 2023. Of the 148 screened participants, 140 were eligible for enrollment and were randomized.
  No participants were enrolled into Cohorts 5, 6, or 7.
Groups:
- Cohort 1 - 9-17 Yrs, 1 Dose 10^9 TCID50 Sing2016 M2SR H3N2; Cohort 3 - 2-8 Yrs, 1 Dose 10^9 TCID50 Sing2016 M2SR H3N2: 10^9 TCID50 of a novel intranasal live attenuated influenza vaccine with a defective M2 gene which renders the virus unable to replicate and generate progeny in animals and in humans, making its infectivity self-limiting. It induces both a mucosal and cell-mediated immune response and is administered intranasally. Supplied by Flugen Inc. One dose administered intranasally on Day 1.
- Cohort 1 - 9-17 Yrs, 1 Dose Placebo; Cohort 2 - 2-8 Yrs, 1 Dose Placebo; Cohort 3 - 2-8 Yrs, 1 Dose Placebo: Physiological saline, i.e., 0.9% sodium chloride. One dose administered intranasally on Day 1.
- Cohort 2 - 2-8 Yrs, 1 Dose 10^8 TCID50 Sing2016 M2SR H3N2: 10^8 TCID50 of a novel intranasal live attenuated influenza vaccine with a defective M2 gene which renders the virus unable to replicate and generate progeny in animals and in humans, making its infectivity self-limiting. It induces both a mucosal and cell-mediated immune response and is administered intranasally. Supplied by Flugen Inc. One dose administered intranasally on Day 1.
- Cohort 4 - 2-8 Yrs, 2 Doses 10^9 TCID50 Sing2016 M2SR H3N2: 10^9 TCID50 of a novel intranasal live attenuated influenza vaccine with a defective M2 gene which renders the virus unable to replicate and generate progeny in animals and in humans, making its infectivity self-limiting. It induces both a mucosal and cell-mediated immune response and is administered intranasally. Supplied by Flugen Inc. Two doses: one administered intranasally on Day 1, and the second administered intranasally on approximately Day 29.
- Cohort 4 - 2-8 Yrs, 2 Doses Placebo: Physiological saline, i.e., 0.9% sodium chloride. Two doses: one administered intranasally on Day 1, and the second administered intranasally on approximately Day 29.
Period: Overall Study
Arm/Group | Cohort 1 - 9-17 Yrs, 1 Dose 10^9 TCID50 Sing2016 M2SR H3N2 | Cohort 1 - 9-17 Yrs, 1 Dose Placebo | Cohort 2 - 2-8 Yrs, 1 Dose 10^8 TCID50 Sing2016 M2SR H3N2 | Cohort 2 - 2-8 Yrs, 1 Dose Placebo | Cohort 3 - 2-8 Yrs, 1 Dose 10^9 TCID50 Sing2016 M2SR H3N2 | Cohort 3 - 2-8 Yrs, 1 Dose Placebo | Cohort 4 - 2-8 Yrs, 2 Doses 10^9 TCID50 Sing2016 M2SR H3N2 | Cohort 4 - 2-8 Yrs, 2 Doses Placebo
Started | 31 | 14 | 30 | 15 | 15 | 10 | 14 | 11
Withdrawal by Subject | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Withdrawal by Parent/Guardian | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Completed | 30 | 14 | 28 | 14 | 15 | 10 | 13 | 11
Not Completed | 1 | 0 | 2 | 1 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1 - 9-17 Yrs, 1 Dose 10^9 TCID50 Sing2016 M2SR H3N2 | Cohort 1 - 9-17 Yrs, 1 Dose Placebo | Cohort 2 - 2-8 Yrs, 1 Dose 10^8 TCID50 Sing2016 M2SR H3N2 | Cohort 2 - 2-8 Yrs, 1 Dose Placebo | Cohort 3 - 2-8 Yrs, 1 Dose 10^9 TCID50 Sing2016 M2SR H3N2 | Cohort 3 - 2-8 Yrs, 1 Dose Placebo | Cohort 4 - 2-8 Yrs, 2 Doses 10^9 TCID50 Sing2016 M2SR H3N2 | Cohort 4 - 2-8 Yrs, 2 Doses Placebo | Total
Number analyzed (Participants) | 31 | 14 | 30 | 15 | 15 | 10 | 14 | 11 | 140
Age, Continuous [Mean (Standard Deviation); unit: years] | 12.5 (2.4) | 13.4 (2.5) | 5.3 (1.6) | 4.3 (2) | 5.7 (2) | 5.4 (2.1) | 5.1 (2.2) | 5.2 (1.8) | 7.6 (4.1)
Age, Customized [Count of Participants; unit: Participants]
  2-4 years old | 0 | 0 | 8 | 8 | 4 | 3 | 5 | 4 | 32
  5-8 years old | 0 | 0 | 22 | 7 | 11 | 7 | 9 | 7 | 63
  9-17 years old | 31 | 14 | 0 | 0 | 0 | 0 | 0 | 0 | 45
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 5 | 15 | 9 | 5 | 3 | 7 | 7 | 67
  Male | 15 | 9 | 15 | 6 | 10 | 7 | 7 | 4 | 73
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 0 | 6 | 0 | 0 | 0 | 1 | 2 | 11
  Not Hispanic or Latino | 29 | 14 | 24 | 15 | 15 | 10 | 13 | 9 | 129
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 2 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 5 | 1 | 2 | 0 | 1 | 1 | 0 | 0 | 10
  White | 22 | 12 | 25 | 14 | 11 | 6 | 11 | 7 | 108
  More than one race | 2 | 1 | 3 | 1 | 2 | 3 | 3 | 4 | 19
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 31 | 14 | 30 | 15 | 15 | 10 | 14 | 11 | 140

OUTCOME MEASURES:

1. Primary Outcome: Number and Percentage of Participants Experiencing a Solicited Reactogenicity Adverse Event
Description: Number and percentage of participants in Cohorts 1-4 each and across Cohorts 1-4 who experience systemic (solicited or local) reactogenicity events, of all severity grades and by grade
Time Frame: Day of first vaccination through 7 days post-dose 1
Population: As pre-specified in Statistical Analysis Plan, vaccine recipients in Cohorts 3&4 are intentionally combined and placebo participants in Cohorts 2-4 are intentionally combined. The safety population consists of all participants who received at least one study influenza vaccination
Measure: Count of Participants; unit: Participants
Groups:
- Cohort 3 & 4 - Vaccine: Cohorts 3 and 4 combined
- Cohort 2, 3, 4 - Placebo: Cohorts 2, 3, and 4 combined
- All Participants - Vaccine: All participants who received vaccine
- All Participants - Placebo: All participants who received Placebo
Arm/Group | Cohort 1 - 9-17 Yrs, 1 Dose 10^9 TCID50 Sing2016 M2SR H3N2 | Cohort 1 - 9-17 Yrs, 1 Dose Placebo | Cohort 2 - 2-8 Yrs, 1 Dose 10^8 TCID50 Sing2016 M2SR H3N2 | Cohort 3 & 4 - Vaccine | Cohort 2, 3, 4 - Placebo | All Participants - Vaccine | All Participants - Placebo
Number analyzed (Participants) | 31 | 14 | 30 | 29 | 36 | 90 | 50
Participants
  Any Solicited Event: None | 14 | 4 | 8 | 8 | 8 | 30 | 12
  Any Solicited Event: Mild | 16 | 5 | 18 | 19 | 23 | 53 | 28
  Any Solicited Event: Moderate | 1 | 5 | 4 | 2 | 5 | 7 | 10
  Any Solicited Event: Severe | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Any Local Solicited Event: None | 21 | 6 | 10 | 10 | 12 | 41 | 18
  Any Local Solicited Event: Mild | 9 | 4 | 16 | 18 | 21 | 43 | 25
  Any Local Solicited Event: Moderate | 1 | 4 | 4 | 1 | 3 | 6 | 7
  Any Local Solicited Event: Severe | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Any Systemic Solicited Event: None | 16 | 6 | 16 | 16 | 17 | 48 | 23
  Any Systemic Solicited Event: Mild | 15 | 5 | 12 | 12 | 14 | 39 | 19
  Any Systemic Solicited Event: Moderate | 0 | 3 | 2 | 1 | 5 | 3 | 8
  Any Systemic Solicited Event: Severe | 0 | 0 | 0 | 0 | 0 | 0 | 0

2. Primary Outcome: Number and Percentage of Participants Experiencing a Solicited Reactogenicity Adverse Event
Description: Number and percentage of participants in Cohort 4 who experience systemic (solicited or local) reactogenicity events, of all severity grades and by grade
Time Frame: Day of second vaccination through 7 days post-dose 2 (Day 29 to Day 36)
Population: The safety population consists of all participants who received at least two study influenza vaccination
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 4 - 2-8 Yrs, 2 Doses 10^9 TCID50 Sing2016 M2SR H3N2 | Cohort 4 - 2-8 Yrs, 2 Doses Placebo
Number analyzed (Participants) | 12 | 11
Participants
  Any Solicited Event: None | 5 | 4
  Any Solicited Event: Mild | 6 | 5
  Any Solicited Event: Moderate | 1 | 0
  Any Solicited Event: Severe | 0 | 2
  Any Local Solicited Event: None | 7 | 6
  Any Local Solicited Event: Mild | 4 | 5
  Any Local Solicited Event: Moderate | 1 | 0
  Any Local Solicited Event: Severe | 0 | 0
  Any Systemic Solicited Event: None | 8 | 5
  Any Systemic Solicited Event: Mild | 4 | 4
  Any Systemic Solicited Event: Moderate | 0 | 0
  Any Systemic Solicited Event: Severe | 0 | 2

3. Primary Outcome: Number and Percentage of Participants Experiencing an Unsolicited Non-serious Adverse Event (AE)
Description: Number and percentage of participants in Cohorts 1-4 each and across Cohorts 1-4 who experience unsolicited non-serious adverse events, of all severity grades and by grade
Time Frame: Day of first vaccination through 28 days post-dose 1
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 - 9-17 Yrs, 1 Dose 10^9 TCID50 Sing2016 M2SR H3N2 | Cohort 1 - 9-17 Yrs, 1 Dose Placebo | Cohort 2 - 2-8 Yrs, 1 Dose 10^8 TCID50 Sing2016 M2SR H3N2 | Cohort 3 & 4 - Vaccine | Cohort 2, 3, 4 - Placebo
Number analyzed (Participants) | 31 | 14 | 30 | 29 | 36
Participants
  Mild | 1 | 3 | 4 | 5 | 3
  Moderate | 1 | 1 | 3 | 0 | 4
  Severe | 0 | 0 | 0 | 0 | 0

4. Primary Outcome: Number and Percentage of Participants Experiencing an Unsolicited Non-serious Adverse Event (AE)
Description: Number and percentage of participants in Cohort 4 who experience unsolicited non-serious adverse events, of all severity grades and by grade
Time Frame: Day of second vaccination through 7 days post-dose 2 (Day 29 to Day 36)
Population: The safety population consists of all participants who received at least two study influenza vaccination
Measure: Count of Participants; unit: Participants
Groups:
- Cohort 4 - 2-8 Yrs, 2 Doses Placebo: 0.9% sodium chloride. Two doses: one administered intranasally on Day 1, and the second administered intranasally on approximately Day 29.
Arm/Group | Cohort 4 - 2-8 Yrs, 2 Doses 10^9 TCID50 Sing2016 M2SR H3N2 | Cohort 4 - 2-8 Yrs, 2 Doses Placebo
Number analyzed (Participants) | 12 | 11
Participants
  Mild | 0 | 2
  Moderate | 1 | 2
  Severe | 0 | 0

5. Primary Outcome: Number and Percentage of Participants Experiencing an Adverse Event of Special Interest (AESI)
Description: Number and percentage of participants in Cohorts 1-4 each and across Cohorts 1-4 who experience AESIs
Time Frame: Day 1 through final visit in the month of April of the calendar year following enrollment (up to 14 months post-baseline)
Population: The safety population consists of all participants who received at least one study influenza vaccination
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 - 9-17 Yrs, 1 Dose 10^9 TCID50 Sing2016 M2SR H3N2 | Cohort 1 - 9-17 Yrs, 1 Dose Placebo | Cohort 2 - 2-8 Yrs, 1 Dose 10^8 TCID50 Sing2016 M2SR H3N2 | Cohort 2 - 2-8 Yrs, 1 Dose Placebo | Cohort 3 - 2-8 Yrs, 1 Dose 10^9 TCID50 Sing2016 M2SR H3N2 | Cohort 3 - 2-8 Yrs, 1 Dose Placebo | Cohort 4 - 2-8 Yrs, 2 Doses 10^9 TCID50 Sing2016 M2SR H3N2 | Cohort 4 - 2-8 Yrs, 2 Doses Placebo
Number analyzed (Participants) | 31 | 14 | 30 | 15 | 15 | 10 | 14 | 11
Participants | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0

6. Primary Outcome: Number and Percentage of Participants Experiencing a Serious Adverse Event (SAE)
Description: Number and percentage of participants in Cohorts 1-4 each and across Cohorts 1-4 who experience serious adverse events (SAEs)
Time Frame: as for outcome 5
Population: The safety population consists of all participants who received at least one study influenza vaccination
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 - 9-17 Yrs, 1 Dose 10^9 TCID50 Sing2016 M2SR H3N2 | Cohort 1 - 9-17 Yrs, 1 Dose Placebo | Cohort 2 - 2-8 Yrs, 1 Dose 10^8 TCID50 Sing2016 M2SR H3N2 | Cohort 2 - 2-8 Yrs, 1 Dose Placebo | Cohort 3 - 2-8 Yrs, 1 Dose 10^9 TCID50 Sing2016 M2SR H3N2 | Cohort 3 - 2-8 Yrs, 1 Dose Placebo | Cohort 4 - 2-8 Yrs, 2 Doses 10^9 TCID50 Sing2016 M2SR H3N2 | Cohort 4 - 2-8 Yrs, 2 Doses Placebo
Number analyzed (Participants) | 31 | 14 | 30 | 15 | 15 | 10 | 14 | 11
Participants | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0

7. Primary Outcome: Number and Percentage of Participants Experiencing a New-onset Chronic Medical Condition (NOCMC)
Description: Number and percentage of participants in Cohorts 1-4 each and across Cohorts 1-4 who experience new-onset chronic medical conditions (NOCMCs)
Time Frame: as for outcome 5
Population: The safety population consists of all participants who received at least one study influenza vaccination
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 - 9-17 Yrs, 1 Dose 10^9 TCID50 Sing2016 M2SR H3N2 | Cohort 1 - 9-17 Yrs, 1 Dose Placebo | Cohort 2 - 2-8 Yrs, 1 Dose 10^8 TCID50 Sing2016 M2SR H3N2 | Cohort 2 - 2-8 Yrs, 1 Dose Placebo | Cohort 3 - 2-8 Yrs, 1 Dose 10^9 TCID50 Sing2016 M2SR H3N2 | Cohort 3 - 2-8 Yrs, 1 Dose Placebo | Cohort 4 - 2-8 Yrs, 2 Doses 10^9 TCID50 Sing2016 M2SR H3N2 | Cohort 4 - 2-8 Yrs, 2 Doses Placebo
Number analyzed (Participants) | 31 | 14 | 30 | 15 | 15 | 10 | 14 | 11
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

8. Secondary Outcome: Number and Percentage of Participants With Putative Seroprotection Against an H3N2 M2SR-like Virus
Description: Titers for each participant are estimated as the geometric mean of technical replicate results. Putative seroprotection is defined as a serum hemagglutination inhibition (HAI) antibody titer greater than or equal to 1:40
Time Frame: Day 1, Day 29 (Cohorts 1, 2, and 3), and Day 57 (Cohort 4)
Population: The modified intent-to-treat population consists of all participants who received study influenza vaccination and had a baseline and at least one post-baseline sample available corresponding to at least one secondary immunogenicity assay
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 - 9-17 Yrs, 1 Dose 10^9 TCID50 Sing2016 M2SR H3N2 | Cohort 1 - 9-17 Yrs, 1 Dose Placebo | Cohort 2 - 2-8 Yrs, 1 Dose 10^8 TCID50 Sing2016 M2SR H3N2 | Cohort 2 - 2-8 Yrs, 1 Dose Placebo | Cohort 3 - 2-8 Yrs, 1 Dose 10^9 TCID50 Sing2016 M2SR H3N2 | Cohort 3 - 2-8 Yrs, 1 Dose Placebo | Cohort 4 - 2-8 Yrs, 2 Doses 10^9 TCID50 Sing2016 M2SR H3N2 | Cohort 4 - 2-8 Yrs, 2 Doses Placebo
Number analyzed (Participants) | 31 | 14 | 29 | 15 | 15 | 10 | 13 | 11
Participants
  Day 1 | 30 | 13 | 16 | 5 | 10 | 6 | 5 | 5
  Day 29 (Cohorts 1, 2, 3): number analyzed (Participants) | 31 | 14 | 29 | 14 | 12 | 9 | 0 | 0
  Day 29 (Cohorts 1, 2, 3) | 30 | 13 | 14 | 4 | 8 | 5 |  |
  Day 57 (Cohort 4): number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 11 | 11
  Day 57 (Cohort 4) |  |  |  |  |  |  | 4 | 5

9. Secondary Outcome: Number and Percentage of Participants With Serum Neutralizing Antibody Titer Against an H3N2 M2SR-like Virus Greater Than or Equal to 1:40
Description: Titers for each participant are estimated as the geometric mean of technical replicate results.
Time Frame: Day 1, Day 29 (Cohorts 1, 2, and 3), and Day 57 (Cohort 4)
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 - 9-17 Yrs, 1 Dose 10^9 TCID50 Sing2016 M2SR H3N2 | Cohort 1 - 9-17 Yrs, 1 Dose Placebo | Cohort 2 - 2-8 Yrs, 1 Dose 10^8 TCID50 Sing2016 M2SR H3N2 | Cohort 2 - 2-8 Yrs, 1 Dose Placebo | Cohort 3 - 2-8 Yrs, 1 Dose 10^9 TCID50 Sing2016 M2SR H3N2 | Cohort 3 - 2-8 Yrs, 1 Dose Placebo | Cohort 4 - 2-8 Yrs, 2 Doses 10^9 TCID50 Sing2016 M2SR H3N2 | Cohort 4 - 2-8 Yrs, 2 Doses Placebo
Number analyzed (Participants) | 31 | 14 | 29 | 15 | 15 | 10 | 13 | 11
Participants
  Day 1 | 31 | 13 | 19 | 9 | 10 | 7 | 6 | 7
  Day 29 (Cohorts 1, 2, 3): number analyzed (Participants) | 31 | 14 | 29 | 14 | 12 | 9 | 0 | 0
  Day 29 (Cohorts 1, 2, 3) | 31 | 13 | 19 | 9 | 9 | 5 |  |
  Day 57 (Cohort 4): number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 11 | 11
  Day 57 (Cohort 4) |  |  |  |  |  |  | 7 | 8

10. Secondary Outcome: Geometric Mean Titers (GMTs) of Serum Hemagglutination Inhibition (HAI) Antibodies Against an H3N2 M2SR-like Virus
Description: Titers for each participant are estimated as the geometric mean of technical replicate results, and the geometric mean is taken again across participants in each group at each time point.
Time Frame: Day 1, Day 29 (Cohorts 1, 2, and 3), and Day 57 (Cohort 4)
Population: as for outcome 8
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Cohort 1 - 9-17 Yrs, 1 Dose 10^9 TCID50 Sing2016 M2SR H3N2 | Cohort 1 - 9-17 Yrs, 1 Dose Placebo | Cohort 2 - 2-8 Yrs, 1 Dose 10^8 TCID50 Sing2016 M2SR H3N2 | Cohort 2 - 2-8 Yrs, 1 Dose Placebo | Cohort 3 - 2-8 Yrs, 1 Dose 10^9 TCID50 Sing2016 M2SR H3N2 | Cohort 3 - 2-8 Yrs, 1 Dose Placebo | Cohort 4 - 2-8 Yrs, 2 Doses 10^9 TCID50 Sing2016 M2SR H3N2 | Cohort 4 - 2-8 Yrs, 2 Doses Placebo
Number analyzed (Participants) | 31 | 14 | 29 | 15 | 15 | 10 | 13 | 11
titer
  Day 1 | 250.2 [178.9 to 342.2] | 190.3 [90.5 to 353.3] | 43 [23.6 to 78.1] | 25.2 [13.8 to 50.4] | 51.6 [23.5 to 113.1] | 60.6 [28.3 to 139.3] | 20 [11.7 to 36] | 28.3 [16 to 54.8]
  Day 29 (Cohorts 1, 2, and 3): number analyzed (Participants) | 31 | 14 | 29 | 14 | 12 | 9 | 0 | 0
  Day 29 (Cohorts 1, 2, and 3) | 242 [171.1 to 334.6] | 119.9 [102.5 to 353.3] | 41 [13.1 to 72.7] | 21 [13.5 to 34.5] | 58.2 [26.7 to 134.5] | 50.4 [20 to 127] |  |
  Day 57 (Cohort 4): number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 11 | 11
  Day 57 (Cohort 4) |  |  |  |  |  |  | 24.9 [14.4 to 44] | 24.9 [13.7 to 46.8]

11. Secondary Outcome: Geometric Mean Titers (GMTs) of Serum Neutralizing Antibodies Against an H3N2 M2SR-like Virus
Description: as for outcome 10
Time Frame: Day 1, Day 29 (Cohorts 1, 2, and 3), and Day 57 (Cohort 4)
Population: as for outcome 8
Measure: Geometric Mean (95% Confidence Interval); unit: titers
Arm/Group | Cohort 1 - 9-17 Yrs, 1 Dose 10^9 TCID50 Sing2016 M2SR H3N2 | Cohort 1 - 9-17 Yrs, 1 Dose Placebo | Cohort 2 - 2-8 Yrs, 1 Dose 10^8 TCID50 Sing2016 M2SR H3N2 | Cohort 2 - 2-8 Yrs, 1 Dose Placebo | Cohort 3 - 2-8 Yrs, 1 Dose 10^9 TCID50 Sing2016 M2SR H3N2 | Cohort 3 - 2-8 Yrs, 1 Dose Placebo | Cohort 4 - 2-8 Yrs, 2 Doses 10^9 TCID50 Sing2016 M2SR H3N2 | Cohort 4 - 2-8 Yrs, 2 Doses Placebo
Number analyzed (Participants) | 31 | 14 | 29 | 15 | 15 | 10 | 13 | 11
titers
  Day 1 | 585.2 [409.2 to 837] | 499.7 [204.9 to 999.3] | 77.2 [39.5 to 154.4] | 45.9 [21.4 to 100.8] | 85.7 [31 to 223.7] | 105.6 [40 to 269.2] | 27.5 [13.1 to 59.7] | 46.8 [20 to 106.2]
  Day 29 (Cohorts 1, 2, 3): number analyzed (Participants) | 31 | 14 | 29 | 14 | 12 | 9 | 0 | 0
  Day 29 (Cohorts 1, 2, 3) | 598.5 [418.5 to 846.4] | 512.2 [210.1 to 1050] | 76.3 [39.5 to 148.9] | 41 [19 to 88.3] | 106.8 [36.7 to 320] | 89.8 [30.5 to 254] |  |
  Day 57 (Cohort 4): number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 11 | 11
  Day 57 (Cohort 4) |  |  |  |  |  |  | 42.6 [20.6 to 85.2] | 53.1 [22.7 to 120.5]

12. Secondary Outcome: Geometric Mean Fold Rise (GMFR) in Serum Hemagglutination Inhibition (HAI) Antibody Titers Against an H3N2 M2SR-like Virus
Description: Titers for each participant are estimated as the geometric mean of technical replicate results. Fold-rise in titers is calculated as the post-vaccination titer divided by the pre-vaccination titer. The geometric mean of fold-rises is taken again across participants in each group at each time point.
Time Frame: Day 29 (Cohorts 1, 2, and 3) and Day 57 (Cohort 4)
Population: as for outcome 8
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | Cohort 1 - 9-17 Yrs, 1 Dose 10^9 TCID50 Sing2016 M2SR H3N2 | Cohort 1 - 9-17 Yrs, 1 Dose Placebo | Cohort 2 - 2-8 Yrs, 1 Dose 10^8 TCID50 Sing2016 M2SR H3N2 | Cohort 2 - 2-8 Yrs, 1 Dose Placebo | Cohort 3 - 2-8 Yrs, 1 Dose 10^9 TCID50 Sing2016 M2SR H3N2 | Cohort 3 - 2-8 Yrs, 1 Dose Placebo | Cohort 4 - 2-8 Yrs, 2 Doses 10^9 TCID50 Sing2016 M2SR H3N2 | Cohort 4 - 2-8 Yrs, 2 Doses Placebo
Number analyzed (Participants) | 31 | 14 | 29 | 15 | 15 | 10 | 13 | 11
Ratio
  Day 29 (Cohorts 1, 2, and 3): number analyzed (Participants) | 31 | 14 | 29 | 14 | 12 | 9 | 0 | 0
  Day 29 (Cohorts 1, 2, and 3) | 1 [.9 to 1.1] | 1.1 [.9 to 1.3] | 1 [.9 to 1.1] | 1 [.8 to 1.2] | 1 [.8 to 1.3] | .9 [.8 to 1] |  |
  Day 57 (Cohort 4): number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 11 | 11
  Day 57 (Cohort 4) |  |  |  |  |  |  | 1.3 [1.1 to 1.8] | .9 [.7 to 1.2]

13. Secondary Outcome: Geometric Mean Fold Rise (GMFR) in Serum Neutralizing Antibody Titers Against an H3N2 M2SR-like Virus
Description: as for outcome 12
Time Frame: Day 29 (Cohorts 1, 2, and 3) and Day 57 (Cohort 4)
Population: as for outcome 8
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | Cohort 1 - 9-17 Yrs, 1 Dose 10^9 TCID50 Sing2016 M2SR H3N2 | Cohort 1 - 9-17 Yrs, 1 Dose Placebo | Cohort 2 - 2-8 Yrs, 1 Dose 10^8 TCID50 Sing2016 M2SR H3N2 | Cohort 2 - 2-8 Yrs, 1 Dose Placebo | Cohort 3 - 2-8 Yrs, 1 Dose 10^9 TCID50 Sing2016 M2SR H3N2 | Cohort 3 - 2-8 Yrs, 1 Dose Placebo | Cohort 4 - 2-8 Yrs, 2 Doses 10^9 TCID50 Sing2016 M2SR H3N2 | Cohort 4 - 2-8 Yrs, 2 Doses Placebo
Number analyzed (Participants) | 31 | 14 | 29 | 15 | 15 | 10 | 13 | 11
Ratio
  Day 29 (Cohorts 1, 2, and 3): number analyzed (Participants) | 31 | 14 | 29 | 14 | 12 | 10 | 0 | 0
  Day 29 (Cohorts 1, 2, and 3) | 1 [.9 to 1.1] | 1 [1 to 1.1] | 1 [.9 to 1.1] | 1.1 [1 to 1.2] | 1.2 [1 to 1.4] | 1 [.8 to 1.1] |  |
  Day 57 (Cohort 4): number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 11 | 11
  Day 57 (Cohort 4) |  |  |  |  |  |  | 1.9 [1.2 to 3.3] | 1.1 [1 to 1.3]

14. Secondary Outcome: Percentage of Participants With Greater Than or Equal to 2- and 4-fold Mean Rises in Hemagglutination Inhibition (HAI) Antibody Titer Against an H3N2 M2SR-like Virus
Description: Titers for each participant are estimated as the geometric mean of technical replicate results. Fold-rise in titers is calculated as the post-vaccination titer divided by the pre-vaccination titer.
Time Frame: Day 29 (Cohorts 1, 2, and 3) and Day 57 (Cohort 4)
Population: as for outcome 8
Measure: Number (95% Confidence Interval); unit: percent of participants
Arm/Group | Cohort 1 - 9-17 Yrs, 1 Dose 10^9 TCID50 Sing2016 M2SR H3N2 | Cohort 1 - 9-17 Yrs, 1 Dose Placebo | Cohort 2 - 2-8 Yrs, 1 Dose 10^8 TCID50 Sing2016 M2SR H3N2 | Cohort 2 - 2-8 Yrs, 1 Dose Placebo | Cohort 3 - 2-8 Yrs, 1 Dose 10^9 TCID50 Sing2016 M2SR H3N2 | Cohort 3 - 2-8 Yrs, 1 Dose Placebo | Cohort 4 - 2-8 Yrs, 2 Doses 10^9 TCID50 Sing2016 M2SR H3N2 | Cohort 4 - 2-8 Yrs, 2 Doses Placebo
Number analyzed (Participants) | 31 | 14 | 29 | 15 | 15 | 10 | 13 | 11
percent of participants
  =>2 Fold-rise Day 29 (Cohorts 1, 2, and 3): number analyzed (Participants) | 31 | 14 | 29 | 14 | 12 | 9 | 0 | 0
  =>2 Fold-rise Day 29 (Cohorts 1, 2, and 3) | 9.7 [2 to 25.8] | 14.3 [1.8 to 42.8] | 6.9 [.8 to 22.8] | 14.3 [1.8 to 42.8] | 16.7 [2.1 to 48.4] | 0 [0 to 33.6] |  |
  =>2 Fold-rise Day 57 (Cohort 4): number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 11 | 11
  =>2 Fold-rise Day 57 (Cohort 4) |  |  |  |  |  |  | 27.3 [6 to 61] | 18.2 [2.3 to 51.8]
  =>4 Fold-rise Day 29 (Cohorts 1, 2, and 3): number analyzed (Participants) | 31 | 14 | 29 | 14 | 12 | 9 | 0 | 0
  =>4 Fold-rise Day 29 (Cohorts 1, 2, and 3) | 0 [0 to 11.2] | 0 [0 to 23.2] | 0 [0 to 11.9] | 0 [0 to 23.2] | 0 [0 to 26.5] | 0 [0 to 33.6] |  |
  =>4 Fold-rise Day 57 (Cohort 4): number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 11 | 11
  =>4 Fold-rise Day 57 (Cohort 4) |  |  |  |  |  |  | 9.1 [.2 to 41.3] | 0 [0 to 28.5]

15. Secondary Outcome: Percent of Participants With Greater Than or Equal to 2- and 4-fold Mean Rises in Serum Neutralizing Antibody Titer Against an H3N2 M2SR-like Virus
Description: as for outcome 14
Time Frame: Day 29 (Cohorts 1, 2, and 3) and Day 57 (Cohort 4)
Population: as for outcome 8
Measure: Number (95% Confidence Interval); unit: percent of participants
Arm/Group | Cohort 1 - 9-17 Yrs, 1 Dose 10^9 TCID50 Sing2016 M2SR H3N2 | Cohort 1 - 9-17 Yrs, 1 Dose Placebo | Cohort 2 - 2-8 Yrs, 1 Dose 10^8 TCID50 Sing2016 M2SR H3N2 | Cohort 2 - 2-8 Yrs, 1 Dose Placebo | Cohort 3 - 2-8 Yrs, 1 Dose 10^9 TCID50 Sing2016 M2SR H3N2 | Cohort 3 - 2-8 Yrs, 1 Dose Placebo | Cohort 4 - 2-8 Yrs, 2 Doses 10^9 TCID50 Sing2016 M2SR H3N2 | Cohort 4 - 2-8 Yrs, 2 Doses Placebo
Number analyzed (Participants) | 31 | 14 | 29 | 15 | 15 | 10 | 13 | 11
percent of participants
  =>2 Fold-rise Day 29 (Cohorts 1, 2, and 3): number analyzed (Participants) | 31 | 14 | 29 | 14 | 12 | 9 | 0 | 0
  =>2 Fold-rise Day 29 (Cohorts 1, 2, and 3) | 6.5 [.8 to 21.4] | 0 [0 to 23.2] | 10.3 [2.2 to 27.4] | 7.1 [.2 to 33.9] | 16.7 [2.1 to 48.4] | 0 [0 to 33.6] |  |
  =>2 Fold-rise Day 57 (Cohort 4): number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 11 | 11
  =>2 Fold-rise Day 57 (Cohort 4) |  |  |  |  |  |  | 27.3 [6 to 61] | 9.1 [.2 to 41.3]
  =>4 Fold-rise Day 29 (Cohorts 1, 2, and 3): number analyzed (Participants) | 31 | 14 | 29 | 15 | 12 | 9 | 0 | 0
  =>4 Fold-rise Day 29 (Cohorts 1, 2, and 3) | 0 [0 to 11.2] | 0 [0 to 23.2] | 0 [0 to 11.9] | 0 [0 to 23.2] | 0 [0 to 26.5] | 0 [0 to 33.6] |  |
  =>4 Fold-rise Day 57 (Cohort 4): number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 11 | 11
  =>4 Fold-rise Day 57 (Cohort 4) |  |  |  |  |  |  | 27.3 [6 to 61] | 0 [0 to 28.5]

16. Secondary Outcome: Mean Secretory Immunoglobulin A (sIgA) Response (i.e., Specific Activity) as Measured by a Binding Antibody Multiplex Assay (BAMA) in Nasal Lavage Specimens Against an H3N2 M2SR-like Virus
Description: Antigen-specific electrochemiluminescence (ECL) signal is calculated as the antigen specific background-subtracted ECL signal times the dilution factor at the replicate level. secretory Immunoglobulin A (sIgA) specific activity is calculated as the arithmetic mean of the antigen-specific ECL signal replicates divided by the arithmetic mean of the total sIgA concentration replicates. The arithmetic mean is taken again across participants in each group at each time point.
  Measured in Mean ECL luminosity signal, as arbitrary units (AU) against each antigen over ug/L sIgA. Higher values correspond to stronger response.
Time Frame: Day 1, Day 29 (Cohorts 1, 2, and 3), and Day 57 (Cohort 4)
Population: as for outcome 8
Measure: Mean (95% Confidence Interval); unit: arbitrary units / ug/L
Arm/Group | Cohort 1 - 9-17 Yrs, 1 Dose 10^9 TCID50 Sing2016 M2SR H3N2 | Cohort 1 - 9-17 Yrs, 1 Dose Placebo | Cohort 2 - 2-8 Yrs, 1 Dose 10^8 TCID50 Sing2016 M2SR H3N2 | Cohort 2 - 2-8 Yrs, 1 Dose Placebo | Cohort 3 - 2-8 Yrs, 1 Dose 10^9 TCID50 Sing2016 M2SR H3N2 | Cohort 3 - 2-8 Yrs, 1 Dose Placebo | Cohort 4 - 2-8 Yrs, 2 Doses 10^9 TCID50 Sing2016 M2SR H3N2 | Cohort 4 - 2-8 Yrs, 2 Doses Placebo
Number analyzed (Participants) | 31 | 14 | 29 | 15 | 15 | 10 | 13 | 11
arbitrary units / ug/L
  Baseline (Texas): number analyzed (Participants) | 31 | 13 | 29 | 15 | 15 | 10 | 13 | 11
  Baseline (Texas) | 2.1 [1.4 to 2.8] | 4.2 [1.4 to 7.9] | 1.8 [.8 to 3.4] | 118.6 [1 to 352.8] | 3.5 [1 to 7.6] | 2.2 [.7 to 4] | 2.1 [1.2 to 3.1] | 2.4 [1.3 to 3.7]
  Day 29 (Texas): number analyzed (Participants) | 31 | 14 | 29 | 15 | 15 | 10 | 0 | 0
  Day 29 (Texas) | 3 [2.1 to 4] | 7.2 [1.8 to 14.5] | 2.2 [.9 to 4] | 1.2 [.9 to 1.7] | 4.5 [1.3 to 8.5] | 9.7 [1.9 to 24] |  |
  Day 57 (Texas): number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 12 | 11
  Day 57 (Texas) |  |  |  |  |  |  | 14.4 [2.6 to 32.8] | 1.9 [.8 to 3.2]
  Baseline (Singapore) | 3.9 [2.3 to 5.7] | 5.4 [2.4 to 9.4] | 3 [1 to 6.1] | 89.3 [1.2 to 263.8] | 6.6 [.7 to 17.9] | 1.4 [.5 to 2.8] | 1.5 [.9 to 2.1] | 2.5 [1.4 to 3.9]
  Day 29 (Singapore): number analyzed (Participants) | 31 | 14 | 29 | 15 | 15 | 10 | 0 | 0
  Day 29 (Singapore) | 6.3 [3.9 to 9.4] | 10.6 [3.8 to 18.9] | 3.7 [1.2 to 7.2] | 1.6 [.8 to 3] | 5.8 [1 to 14] | 1.8 [.5 to 3.3] |  |
  Day 57 (Singapore): number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 12 | 11
  Day 57 (Singapore) |  |  |  |  |  |  | 21.3 [3.3 to 49.4] | 1.8 [.7 to 3.5]
  Baseline (HongKong) | 1.4 [1 to 2] | 1.6 [.9 to 2.5] | 1.2 [.7 to 1.9] | 175.4 [1 to 523.7] | 1.9 [.6 to 3.8] | .9 [.6 to 1.2] | 1.3 [.8 to 1.7] | 2.3 [1 to 4.3]
  Day 29 (HongKong): number analyzed (Participants) | 31 | 14 | 29 | 15 | 15 | 10 | 0 | 0
  Day 29 (HongKong) | 2 [1.4 to 2.6] | 2.6 [.9 to 5.3] | 1.5 [.8 to 2.4] | 1.1 [.7 to 1.6] | 2.2 [1 to 3.8] | 8.6 [1.3 to 22.1] |  |
  Day 57 (HongKong): number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 12 | 11
  Day 57 (HongKong) |  |  |  |  |  |  | 8.4 [1.9 to 18.2] | 1.9 [.7 to 3.5]
  Baseline (Cambodia) | 2 [1.3 to 3] | 2.6 [1.1 to 4.5] | 1.6 [.9 to 2.8] | 133.2 [1.3 to 395.1] | 3.3 [.7 to 8.1] | 2.1 [.8 to 4.2] | 1.7 [1.1 to 2.3] | 1.8 [1 to 2.7]
  Day 29 (Cambodia): number analyzed (Participants) | 31 | 14 | 29 | 15 | 15 | 10 | 0 | 0
  Day 29 (Cambodia) | 2.7 [1.8 to 3.7] | 5 [1.3 to 10.7] | 2.1 [1 to 3.5] | 1.7 [.9 to 3] | 3.3 [1.2 to 6.7] | 4.8 [1.4 to 11] |  |
  Day 57 (Cambodia): number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 12 | 11
  Day 57 (Cambodia) |  |  |  |  |  |  | 15.3 [2 to 38.2] | 1.4 [.7 to 2.6]

17. Secondary Outcome: Mean Change (Difference) From Baseline of Secretory Immunoglobulin A (sIgA) Response (i.e., Specific Activity) as Measured by a Binding Antibody Multiplex Assay (BAMA) in Nasal Lavage Specimens Against an H3N2 M2SR-like Virus
Description: Antigen-specific electrochemiluminescence (ECL) signal is calculated as the antigen specific background-subtracted ECL signal times the dilution factor at the replicate level. secretory Immunoglobulin A (sIgA) specific activity is calculated as the arithmetic mean of the antigen-specific ECL signal replicates divided by the arithmetic mean of the total sIgA concentration replicates. The change from baseline is calculated as the post-vaccination response minus the pre-vaccination response. The arithmetic mean of change from baseline is taken again across participants in each group at each time point.
  Measured in Mean Difference from Baseline in ECL Signal (arbitrary luminescence units) against each antigen over ug/L sIgA. Higher signal represents increased response.
Time Frame: Day 29 (Cohorts 1, 2, and 3) and Day 57 (Cohort 4)
Population: as for outcome 8
Measure: Mean (95% Confidence Interval); unit: arbitrary luminescence units / ug/L
Arm/Group | Cohort 1 - 9-17 Yrs, 1 Dose 10^9 TCID50 Sing2016 M2SR H3N2 | Cohort 1 - 9-17 Yrs, 1 Dose Placebo | Cohort 2 - 2-8 Yrs, 1 Dose 10^8 TCID50 Sing2016 M2SR H3N2 | Cohort 2 - 2-8 Yrs, 1 Dose Placebo | Cohort 3 - 2-8 Yrs, 1 Dose 10^9 TCID50 Sing2016 M2SR H3N2 | Cohort 3 - 2-8 Yrs, 1 Dose Placebo | Cohort 4 - 2-8 Yrs, 2 Doses 10^9 TCID50 Sing2016 M2SR H3N2 | Cohort 4 - 2-8 Yrs, 2 Doses Placebo
Number analyzed (Participants) | 31 | 14 | 29 | 15 | 15 | 10 | 13 | 11
arbitrary luminescence units / ug/L
  Day 29 (Texas): number analyzed (Participants) | 31 | 14 | 29 | 15 | 15 | 10 | 0 | 0
  Day 29 (Texas) | 1 [.3 to 1.8] | 3.5 [0 to 10.3] | .4 [-.1 to 1.1] | -117.4 [-351.8 to .3] | 1.1 [-.9 to 3.4] | 7.6 [.4 to 21] |  |
  Day 57 (Texas): number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 12 | 11
  Day 57 (Texas) |  |  |  |  |  |  | 12.4 [1.1 to 29.9] | -.5 [-1.1 to 0]
  Day 29 (Singapore): number analyzed (Participants) | 31 | 14 | 29 | 15 | 15 | 10 | 0 | 0
  Day 29 (Singapore) | 2.4 [.6 to 4.8] | 5.2 [.3 to 12.9] | .7 [-.1 to 1.8] | -87.7 [-262.1 to .3] | -.9 [-5.1 to 2] | .3 [-1 to 1.6] |  |
  Day 57 (Singapore): number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 12 | 11
  Day 57 (Singapore) |  |  |  |  |  |  | 19.8 [1.7 to 47.6] | -.7 [-1.6 to .1]
  Day 29 (HongKong): number analyzed (Participants) | 31 | 14 | 29 | 15 | 15 | 10 | 0 | 0
  Day 29 (HongKong) | .5 [0 to 1] | 1 [-.7 to 3.7] | .3 [-.1 to .8] | -174.3 [-522.7 to .2] | .4 [-.3 to 1] | 7.7 [.4 to 21] |  |
  Day 57 (HongKong): number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 12 | 11
  Day 57 (HongKong) |  |  |  |  |  |  | 7.1 [.8 to 16.7] | -.4 [-1.1 to .1]
  Day 29 (Cambodia): number analyzed (Participants) | 31 | 14 | 29 | 15 | 15 | 10 | 0 | 0
  Day 29 (Cambodia) | .6 [-.1 to 1.4] | 2.4 [-.4 to 7.5] | .4 [0 to 1.1] | -131.4 [-393 to 0] | -.1 [-1.8 to 1.1] | 2.7 [.2 to 7] |  |
  Day 57 (Cambodia): number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 12 | 11
  Day 57 (Cambodia) |  |  |  |  |  |  | 13.6 [.6 to 36.7] | -.3 [-.6 to 0]

ADVERSE EVENTS:
Time Frame: Solicited AEs collected days 1-8 for all cohorts, days 29-36 for cohort 4. Non-serious, unsolicited AEs collected Days 1-29 for all Cohorts, days 29-57 for Cohort 4. Serious AEs, AEs of special interest, new-onset chronic medical conditions, and all-cause mortality collected up to 14 months post baseline.
Arm/Group | Cohort 1 - 9-17 Yrs, 1 Dose 10^9 TCID50 Sing2016 M2SR H3N2 | Cohort 1 - 9-17 Yrs, 1 Dose Placebo | Cohort 2 - 2-8 Yrs, 1 Dose 10^8 TCID50 Sing2016 M2SR H3N2 | Cohort 2 - 2-8 Yrs, 1 Dose Placebo | Cohort 3 - 2-8 Yrs, 1 Dose 10^9 TCID50 Sing2016 M2SR H3N2 | Cohort 3 - 2-8 Yrs, 1 Dose Placebo | Cohort 4 - 2-8 Yrs, 2 Doses 10^9 TCID50 Sing2016 M2SR H3N2 | Cohort 4 - 2-8 Yrs, 2 Doses Placebo
All-Cause Mortality (participants affected / at risk) | 0/31 | 0/14 | 0/30 | 0/15 | 0/15 | 0/10 | 0/14 | 0/11
Serious Adverse Events (participants affected / at risk) | 0/31 | 0/14 | 0/30 | 0/15 | 1/15 | 0/10 | 0/14 | 0/11
Other Adverse Events (participants affected / at risk) | 17/31 | 10/14 | 22/30 | 11/15 | 12/15 | 9/10 | 12/14 | 8/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 - 9-17 Yrs, 1 Dose 10^9 TCID50 Sing2016 M2SR H3N2 (N=31) | Cohort 1 - 9-17 Yrs, 1 Dose Placebo (N=14) | Cohort 2 - 2-8 Yrs, 1 Dose 10^8 TCID50 Sing2016 M2SR H3N2 (N=30) | Cohort 2 - 2-8 Yrs, 1 Dose Placebo (N=15) | Cohort 3 - 2-8 Yrs, 1 Dose 10^9 TCID50 Sing2016 M2SR H3N2 (N=15) | Cohort 3 - 2-8 Yrs, 1 Dose Placebo (N=10) | Cohort 4 - 2-8 Yrs, 2 Doses 10^9 TCID50 Sing2016 M2SR H3N2 (N=14) | Cohort 4 - 2-8 Yrs, 2 Doses Placebo (N=11)
Pharyngitis (Infections and infestations) | NA | NA | NA | NA | 1 (1) | NA | NA | NA
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 - 9-17 Yrs, 1 Dose 10^9 TCID50 Sing2016 M2SR H3N2 (N=31) | Cohort 1 - 9-17 Yrs, 1 Dose Placebo (N=14) | Cohort 2 - 2-8 Yrs, 1 Dose 10^8 TCID50 Sing2016 M2SR H3N2 (N=30) | Cohort 2 - 2-8 Yrs, 1 Dose Placebo (N=15) | Cohort 3 - 2-8 Yrs, 1 Dose 10^9 TCID50 Sing2016 M2SR H3N2 (N=15) | Cohort 3 - 2-8 Yrs, 1 Dose Placebo (N=10) | Cohort 4 - 2-8 Yrs, 2 Doses 10^9 TCID50 Sing2016 M2SR H3N2 (N=14) | Cohort 4 - 2-8 Yrs, 2 Doses Placebo (N=11)
Eye pruritus (Eye disorders) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Lacrimation increased (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 4 (4) | 1 (1) | 0 (0) | 2 (2) | 3 (3) | 0 (0) | 2 (2) | 2 (2)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 3 (3) | 0 (0) | 3 (3) | 1 (1) | 2 (2) | 1 (1) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 3 (3) | 3 (3) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 2 (2)
Toothache (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Decreased activity (General disorders) | 1 (1) | 3 (3) | 4 (4) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Fatigue (General disorders) | 9 (9) | 5 (5) | 5 (5) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 4 (4)
Malaise (General disorders) | 4 (4) | 4 (4) | 4 (4) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 2 (2)
Pyrexia (General disorders) | 1 (1) | 1 (2) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 4 (9)
COVID-19 (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Otitis media (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Otitis media acute (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pharyngitis streptococcal (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Respiratory syncytial virus infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 2 (2)
Muscle injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 2 (2) | 1 (1) | 5 (5) | 3 (3) | 1 (1) | 1 (1) | 0 (0) | 3 (3)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Headache (Nervous system disorders) | 9 (9) | 5 (5) | 2 (2) | 1 (1) | 4 (4) | 1 (1) | 2 (2) | 2 (2)
Somnolence (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Irritability (Psychiatric disorders) | 0 (0) | 0 (0) | 2 (2) | 3 (3) | 1 (1) | 0 (0) | 3 (3) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 5 (5) | 6 (6) | 6 (6) | 6 (6) | 3 (3) | 6 (7) | 3 (3)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 3 (3) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 8 (8) | 5 (5) | 9 (9) | 4 (4) | 6 (6) | 6 (6) | 6 (7) | 4 (5)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 2 (2) | 3 (3) | 2 (2) | 2 (2) | 1 (1) | 1 (1) | 2 (2)
Paranasal sinus discomfort (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rhinalgia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 3 (3) | 1 (1) | 0 (0) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 6 (6) | 13 (13) | 6 (6) | 9 (9) | 4 (4) | 4 (5) | 3 (3)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 5 (5) | 9 (9) | 2 (2) | 2 (2) | 2 (2) | 3 (3) | 5 (5)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Flushing (Vascular disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eye pruritus (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (3):
  • Study Protocol (2023-12-06): https://cdn.clinicaltrials.gov/large-docs/97/NCT04960397/Prot_001.pdf
  • Statistical Analysis Plan (2024-08-13): https://cdn.clinicaltrials.gov/large-docs/97/NCT04960397/SAP_002.pdf
  • Informed Consent Form (2022-09-26): https://cdn.clinicaltrials.gov/large-docs/97/NCT04960397/ICF_000.pdf